CLINICAL TRIAL: NCT05514145
Title: The Effectiveness of Combined Design Nance/Transpalatal Arch Appliance in Maintaining Arch Dimensions After Premature Extraction of Primary Molars (Randomized Controlled Clinical Trial)
Brief Title: The Effectiveness of Combined Design Nance/Transpalatal Arch Appliance in Maintaining Arch Dimensions After Premature Extraction of Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Elsayed, MSc student, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 301015
Record Dates: First submitted 2022-08-20; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Space Maintenance
Keywords: Nance/transpalatal arch; Nance space maintainer; Space maintainer; Space maintenance

STUDY DESIGN:
Intervention Model Description: Randomized parallel controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nance space maintainer (Active Comparator): Conventional space maintainer for the maxillary arch as control
  Interventions: Device: Nance space maintainer
- Nance/Transpalatal arch space maintainer (Experimental): New design of a space maintainer for the maxillary arch
  Interventions: Device: Nance/Transpalatal arch space maintainer

INTERVENTIONS:
Device: Nance/Transpalatal arch space maintainer — A combined design of both Nance and Transpalatal arch space maintainers as a space maintainer for the maxillary arch in mixed dentition
  Arms: Nance/Transpalatal arch space maintainer
Device: Nance space maintainer — Conventional space maintainer for the maxillary arch used in mixed dentition
  Arms: Nance space maintainer

SUMMARY:
This study will evaluate the effectiveness of N-TPA appliance compared to Nance SM in maintaining the arch dimensions after bilateral premature extraction of primary molars in children.

DETAILED DESCRIPTION:
In this randomized controlled clinical trial, 30 healthy children, 8-9 years of age with premature extraction of bilateral maxillary primary molars will be selected. Children will be randomly allocated into two equal groups of 15 children each according to the type of the appliance that will be used. Group I will receive a a Nance SM, and Group II a combined N-TPA appliance . Panoramic X-rays and study casts will be made, and baseline measurements will be recorded including arch circumference, intermolar width and arch depth. The appliances will be fabricated and cemented intra-orally.

The patients will be followed up at 3, 6 and 9 months for re-evaluation of arch circumference, intermolar width, arch depth, and patient acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Fully erupted maxillary permanent first molars.
* Angle's class I occlusion.(31)
* Adequate space for premolar eruption according to Moyer's arch length analysis.(31)
* Fair to good oral hygiene according to Silness and Loe plaque index.(32)
* No history of allergy to polymethyl methacrylate.

Exclusion Criteria:

* Children with congenitally absent permanent successors.
* Children with successors not covered by bone with 2/3 of the root formed.(33)

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Efficacy in maintaining arch dimensions | 9 months
  All arch dimensions are measured with a 0.5 mm stainless steel wire on the study casts which was then measured with a digital caliper in millimeters (accuracy up to 0.02mm):
  * Changes in arch circumference after insertion of both Nance and Nance/transpalatal arch (N-TPA) appliances after 3, 6- and 9-months follow-up.
  * Changes in intermolar width after insertion of both Nance and Nance/transpalatal arch (N-TPA) appliances after 3, 6- and 9-months follow-up.
  * Changes in arch depth after insertion of both Nance and Nance/transpalatal arch (N-TPA) appliances after 3, 6- and 9-months follow-up.

SECONDARY OUTCOMES:
Patient acceptance by modified faces pain scale | 9 months
  Patient acceptance are measured by the modified faces pain scale of both Nance and N-TPA appliances after 3, 6- and 9-months follow-up.
  Patient acceptance is measured as : (a) Satisfied (b) Indifferent (c) Dissatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No